CLINICAL TRIAL: NCT03536091
Title: Magnification Endoscopy and Electronic Chromoendoscopy in Patients With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Timo Rath, Professor of Endoscopy and Molecular Imaging, University of Erlangen-Nürnberg Medical School
Other Study IDs: EREN IBD
Record Dates: First submitted 2018-05-07; First posted 2018-05-24 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnification endoscopy — All IBD patients will undergo magnification endoscopy with 136-fold optical magnification in conjunction with optical chromoendoscopy

SUMMARY:
In this study the investigators aim to evaluate the ability of i-scan OE together with magnification endoscopy to detect and assess microscopic inflammation in patients with inflammator bowel diseases (IBD).

DETAILED DESCRIPTION:
In this study the investigators aim to evaluate the ability of i-scan OE together with magnification endoscopy to detect and assess microscopic inflammation in patients with inflammator bowel diseases. For this purpose, IBD patients will be prospectively enrolled and inflammatory changes will be assessed using optical magnification endoscopy in conjunction with optical chromoendoscopy. Endoscopic scoring of inflammatory changes in IBD patients will be done on a newly developed magnification score resulting as a consensus from experts in optical diagnosis and endoscopy in IBD patients. Results will be correlated against histopathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established diagnosis of Inflammatory Bowel Diseases
* Ability to provide written informed consent
* Age 18 years and older

Exclusion Criteria:

* poor bowel preparation
* inability to provide written informed consent
* minors

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients treated in the outpatient department of the University Hospital Erlangen
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Assessment of endoscopic Inflammation | 12 months
  Endoscopic Inflammation will be determined and scored by assessement of the vascular and mucosal pattern under magnification endoscopy.
Assessment of histopathological Inflammation | 12 months
  Histopathologic Inflammation will be assessed by grading inflammation of intestinal biopsies routinely obtained during colonoscopy on established pathological scores.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No